CLINICAL TRIAL: NCT03407248
Title: What Are the Roles of Dairy Products in Sustainable Diets? Modelling Nutritional Adequacy, Financial and Environmental Impacts
Brief Title: Dairy Product Consumption and Impact on Nutritional Adequacy, Environment and Diet Cost
Status: Completed | Type: Observational
Sponsor: University of Reading (Other)
Collaborators: Dairy Council, United Kingdom (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Other Study IDs: JAL04
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Diet Pattern Analysis; Environmental Impact; Nutrient Intakes; Cardio-metabolic Health; Dietary Cost

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a secondary analysis of dietary, demographic and health parameter data collected in the 2008/09-2011/12 National Diet and Nutrition Survey (NDNS), UK to determine the roles of dairy products in sustainable diets by modelling nutritional adequacy, financial cost and environmental impact of UK diets containing varying amounts of dairy products.

ELIGIBILITY:
Inclusion Criteria:

* Eligible respondents were adults aged 19-64 years.

Exclusion Criteria:

* Younger than age 18 or older than age 65

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The data included food consumption and nutritional data for 1655 adults (males: n=710 and females: n=945) aged 19-64 years old, in 2008/09-2011/12 National Diet and Nutrition Survey (NDNS).
Sampling Method: Probability Sample
Enrollment: 1655 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Food intake | 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Access to the primary data is available through application to http://www.data-archive.ac.uk

REFERENCES:
- [Derived] Hobbs DA, Durrant C, Elliott J, Givens DI, Lovegrove JA. Diets containing the highest levels of dairy products are associated with greater eutrophication potential but higher nutrient intakes and lower financial cost in the United Kingdom. Eur J Nutr. 2020 Apr;59(3):895-908. doi: 10.1007/s00394-019-01949-y. Epub 2019 Mar 29. PMID 30927064